CLINICAL TRIAL: NCT03079739
Title: The Prospective Assessment of Long-term Outcome of Deferred Coronary Lesions Based on FFR Evaluation
Brief Title: Long-term Outcome of Deferred Lesion Based on FFR
Acronym: HALE-BOPP
Status: Completed | Type: Observational
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Gianluca Campo, Associate Professor, University Hospital of Ferrara
Other Study IDs: 161082
Record Dates: First submitted 2017-03-08; First posted 2017-03-14 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2022-09

CONDITIONS: Myocardial Ischemia
MeSH Terms: conditions — Myocardial Ischemia | interventions — Fractional Flow Reserve, Myocardial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- fractional flow reserve group: consecutive patients undergoing coronary artery angiography for established or suspected ischemic heart disease and receiving in at least one lesion FFR assessment
  Interventions: Diagnostic Test: fractional flow reserve

INTERVENTIONS:
Diagnostic Test: fractional flow reserve — assessment with FFR in at least one coronary lesion

SUMMARY:
Treatment of ischemic myocardium with percutaneous coronary intervention (PCI) in addition to optimal medical therapy reduces major adverse cardiac events. However, less than half of patients have a noninvasive ischemic evaluation before revascularization. Fractional flow reserve (FFR) can determine the hemodynamic significance of a coronary lesion by measuring the distal mean coronary and aortic pressures during maximal hyperemia. Previous studies conducted principally in stable coronary artery disease (CAD) patients have demonstrated that FFR-guided revascularization improves clinical outcomes, quality of life, and cost-efficiency. However, the reliability and safety of FFR assessment in different setting than stable CAD is unclear. In addition, the majority of studies are performed with the only one device. No data are available from other clinically used devices. The HALE BOPP registry is an investigator-initiated observational study, designed to prospectively include all patients referred for coronary angiography in which at least 1 lesion was evaluated by FFR.

DETAILED DESCRIPTION:
Treatment of ischemic myocardium with percutaneous coronary intervention (PCI) in addition to optimal medical therapy reduces major adverse cardiac events. However, less than half of patients have a noninvasive ischemic evaluation before revascularization. Fractional flow reserve (FFR) can determine the hemodynamic significance of a coronary lesion by measuring the distal mean coronary and aortic pressures during maximal hyperemia. Previous studies conducted principally in stable coronary artery disease (CAD) patients have demonstrated that FFR-guided revascularization improves clinical outcomes, quality of life, and cost-efficiency. However, the reliability and safety of FFR assessment in different setting than stable CAD is unclear. In addition, the majority of studies are performed with the only one device. No data are available from other clinically used devices.

The HALE BOPP registry is an investigator-initiated observational study, designed to prospectively include all patients referred for coronary angiography in which at least 1 lesion was evaluated by FFR.

All centers capable of performing FFR were invited to participate and there were no predefined exclusion criteria, other than the patient's unwillingness to provide written informed consent.

The decision to perform FFR was left to the operator in each case. The study primary purpose was to evaluate, in the routine daily practice, the long-term clinical outcome of coronary lesions where the treatment was deferred based on FFR result.

An independent corelab will review all angiograms to perform quantitative coronary analysis, calculation of syntax score, residual syntax score, functional syntax score and, in ACS patients, discrimination between culprit and non culprit lesions An indipendent committee will assess and adjudicate all adverse events.

ELIGIBILITY:
Inclusion Criteria:

* written consent
* age >18 years
* FFR assessment in at least one coronary lesion

Exclusion Criteria:

* life expectancy <1 year because of known noncardiovascular comorbidity
* unwillingness to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients with established or suspected ischemic heart disease referred for coronary artery angiography in which at least 1 lesion is evaluated by FFR.
Sampling Method: Non-Probability Sample
Enrollment: 1305 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
target vessel failure | 1 year
  cumulative occurrence of cardiac death, target vessel myocardial infarction and ischemia-driven target vessel revascularization. The vessel is defined target if it was that where fractional flow reserve is performed.

SECONDARY OUTCOMES:
target vessel failure | 3 years
  cumulative occurrence of cardiac death, target vessel myocardial infarction and ischemia-driven target vessel revascularization. The vessel is defined target if it was that where fractional flow reserve is performed.
target vessel failure | 5 years
  cumulative occurrence of cardiac death, target vessel myocardial infarction and ischemia-driven target vessel revascularization. The vessel is defined target if it was that where fractional flow reserve is performed.

CONTACTS AND LOCATIONS:
Locations (8):
- Italy (8):
  - Clinica Montevergine SPA, Mercogliano, Avellino
  - Istituto Clinico Sant'Anna, Brescia, Brescia
  - Ospedale Valduce, Como, Como
  - University Hospital of Ferrara, Cona, Ferrara
  - Clinica Sant'Ambrogio, Milan, Milano
  - Istituto Auxologico Italiano, Milan, Milano
  - Clinica San Carlo, Paderno Dugnano, Milano
  - AOU di Sassari, Sassari, Sassari

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tebaldi M, Gallo F, Scoccia A, Durante A, Tedeschi D, Verdoliva S, Cortese B, Bilotta F, Watkins S, Ielasi A, Valentini G, Pavasini R, Serenelli M, D'Aniello E, Arena M, Pompei G, Scala A, Scollo E, Gibiino F, Caglioni S, Mele D, Marrone A, Biscaglia S, Barbato E, Campo G. Clinical Outcome of FFR-Guided Revascularization Strategy of Coronary Lesions: The HALE-BOPP Study. Rev Cardiovasc Med. 2023 Feb 14;24(2):62. doi: 10.31083/j.rcm2402062. eCollection 2023 Feb. PMID 39077421